CLINICAL TRIAL: NCT05885815
Title: Application of Surface-enhanced Raman Scatting (SERS) Technology in Clinical Diagnosis and Prognosis of Lung Cancer Immunotherapy
Brief Title: Application of SERS Technology in Clinical Diagnosis and Prognosis of Lung Cancer Immunotherapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Yayi He, Principal Investigator, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 2023HY0520
Record Dates: First submitted 2023-05-20; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Lung Cancer
Keywords: SERS; probes; biopsy; immunotherapy; prognosis
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to explore the application of surface-enhanced Raman scattering (SERS) technology and specific PD-L1 detection fluorescent probes in the clinical diagnosis and prognosis of lung cancer immunotherapy, and further promote the rapid diagnosis of lung cancer and the precision of tumor immunotherapy.

DETAILED DESCRIPTION:
The aim of this study is to explore the application of surface-enhanced Raman scattering (SERS) system in the diagnosis of benign and malignant lung cancer biopsy, and to promote the rapid diagnosis of lung cancer. In addition, the correlation between tumor PH value, PD-L1 expression detected by fluorescent probes and the efficacy and prognosis of immunotherapy was explored. Based on this, the immunotherapy efficacy and prognosis prediction models based on patients' clinical information, PD-L1 expression by immunohistochemistry, PD-L1 expression by fluorescent probes and PH value detected by SERS were constructed to promote the precision of tumor immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in clinical research; Fully understand and informed the study and sign the informed consent form (ICF); Be willing to follow and be able to complete all trial procedures.
2. Male or female aged 18-75 years or more when signing ICF.
3. Fiberoptic bronchoscopy or percutaneous lung biopsy was performed.
4. Lung cancer cannot be surgically resected.
5. At least one measurable target lesion assessed by IRRC according to RECIST 1.1. Patients must provide eligible tumor tissue for PD-L1 expression and PH measurement.

(7) Related laboratory tests suggested that chemotherapy and immunotherapy could be tolerated.

Exclusion Criteria:

1. NSCLC patients with unclear diagnosis;
2. Patients with contraindications to chemotherapy or immunotherapy.
3. Contraindication of lung biopsy.
4. Other active malignant tumors within the past year or at the same time.
5. The patient had a known history of psychotropic drug abuse or drug use; She had a history of alcohol abuse.
6. According to the investigator's judgment, the patient had other factors that may lead to early termination of the study.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Biopsy patients in Shanghai Pulmonary Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
OS | From date of diagnosis until the date of death from any cause, whichever came first, assessed up to 24 months
  Time from randomization to death (from any cause).
PFS | From date of diagnosis until the date of first documented progression from any cause, whichever came first, assessed up to 24 months
  The time between the initiation of randomization and the occurrence (any aspect) of tumor progression or death (from any cause).
ORR | The proportion of patients who achieved a 30%(usual) reduction in tumor volume while maintaining the minimum required duration was calculated at month 24 of the study
  Refers to the proportion of subjects whose tumors shrink by a certain amount and remain for a certain period of time, including those with CR+PR.
DOR | The time from first diagnosis of CR or PR to diagnosis of PD was calculated at 24 months of study.
  Is the time from the first documented response (CR or PR) to the first documented disease progression or death, whichever occurs first.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kennedy LB, Salama AKS. A review of cancer immunotherapy toxicity. CA Cancer J Clin. 2020 Mar;70(2):86-104. doi: 10.3322/caac.21596. Epub 2020 Jan 16. PMID 31944278
- [Result] Postow MA, Callahan MK, Wolchok JD. Immune Checkpoint Blockade in Cancer Therapy. J Clin Oncol. 2015 Jun 10;33(17):1974-82. doi: 10.1200/JCO.2014.59.4358. Epub 2015 Jan 20. PMID 25605845
- [Result] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Result] Hirsch FR, Scagliotti GV, Mulshine JL, Kwon R, Curran WJ Jr, Wu YL, Paz-Ares L. Lung cancer: current therapies and new targeted treatments. Lancet. 2017 Jan 21;389(10066):299-311. doi: 10.1016/S0140-6736(16)30958-8. Epub 2016 Aug 27. PMID 27574741
- [Result] Garon EB, Hellmann MD, Rizvi NA, Carcereny E, Leighl NB, Ahn MJ, Eder JP, Balmanoukian AS, Aggarwal C, Horn L, Patnaik A, Gubens M, Ramalingam SS, Felip E, Goldman JW, Scalzo C, Jensen E, Kush DA, Hui R. Five-Year Overall Survival for Patients With Advanced Non-Small-Cell Lung Cancer Treated With Pembrolizumab: Results From the Phase I KEYNOTE-001 Study. J Clin Oncol. 2019 Oct 1;37(28):2518-2527. doi: 10.1200/JCO.19.00934. Epub 2019 Jun 2. PMID 31154919
- [Result] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leal TA, Riess JW, Jensen E, Zhao B, Pietanza MC, Brahmer JR. Five-Year Outcomes With Pembrolizumab Versus Chemotherapy for Metastatic Non-Small-Cell Lung Cancer With PD-L1 Tumor Proportion Score >/= 50. J Clin Oncol. 2021 Jul 20;39(21):2339-2349. doi: 10.1200/JCO.21.00174. Epub 2021 Apr 19. PMID 33872070
- [Result] Kazdal D, Endris V, Allgauer M, Kriegsmann M, Leichsenring J, Volckmar AL, Harms A, Kirchner M, Kriegsmann K, Neumann O, Brandt R, Talla SB, Rempel E, Ploeger C, von Winterfeld M, Christopoulos P, Merino DM, Stewart M, Allen J, Bischoff H, Meister M, Muley T, Herth F, Penzel R, Warth A, Winter H, Frohling S, Peters S, Swanton C, Thomas M, Schirmacher P, Budczies J, Stenzinger A. Spatial and Temporal Heterogeneity of Panel-Based Tumor Mutational Burden in Pulmonary Adenocarcinoma: Separating Biology From Technical Artifacts. J Thorac Oncol. 2019 Nov;14(11):1935-1947. doi: 10.1016/j.jtho.2019.07.006. Epub 2019 Jul 23. PMID 31349062